CLINICAL TRIAL: NCT02684149
Title: Pain Impact Assessment of the Relational Touch During Arterial Puncture in ICU - TORREA
Brief Title: Pain Impact Assessment of the Relational Touch During Arterial Puncture in ICU (TORREA)
Acronym: ToRRéa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-A01607-40
Record Dates: First submitted 2015-01-21; First posted 2016-02-17 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Pain
Keywords: Intensive care; Arterial puncture; Cross-over; Relational touch; Pain
MeSH Terms: conditions — Pain

ARMS (2):
- A (Experimental): Relational touch before the first arterial puncture and the second arterial puncture without relational touch
  Interventions: Procedure: relational touch
- B (Experimental): First arterial puncture without relational touch and relational touch before the second arterial puncture
  Interventions: Procedure: relational touch

INTERVENTIONS:
Procedure: relational touch

SUMMARY:
Study objective is to assess the interest of the relational touch before an arterial puncture to reduce pain on patient in intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Admission in Intensive Care Unit
* Communicating patient (able to rate their pain on a numerical scale)
* Need for a radial arterial puncture for conducting blood tests, apart for the emergency
* Non-opposition of the patient

Exclusion Criteria:

* Age under 18
* Tetraplegic patient or having a sensitivity disorder on the limb to be punctured
* No radial pulse perception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the variation in pain score (evaluation on a numerical scale 0 to 10) between the measurement made before the arterial puncture and during the arterial puncture. | 1 day
  At the first and second arterial puncture

SECONDARY OUTCOMES:
The change in consumption of analgesics and hypnotics | 1 day
  At the first and second arterial puncture
Blood pressure and heart rate variation | 1 day
  At the first and second arterial puncture
Patient satisfaction score | 1 day
  At the first and second arterial puncture
Number of arterial punctures needed before success | 1 day
  At the first and second arterial puncture

CONTACTS AND LOCATIONS:
Overall Officials: Régine MONCHO, Nurse, Principal Investigator — University Hospital, Angers
Locations (2):
- France (2):
  - University Hospital, Angers
  - University Hospital TOURS, Tours